CLINICAL TRIAL: NCT00309270
Title: A Prospective, Randomized Study to Compare the Effect of Campath-1,Low Dose Sirolimus Versus Campath-1H, Low Dose CsA Both in Addition to Low Dose Mycophenolate Mofetil on Phenotypic and Functional Profiles of PBMCs in Kidney Transplant Recipients in a Steroid-Free Regimen
Brief Title: Low Dose Sirolimus or CsA-Based Maintenance Immunosuppression After Induction With Campath-1 in Kidney Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAMPATH
Record Dates: First submitted 2006-03-30; First posted 2006-03-31 (Estimated); Last update posted 2006-05-22 (Estimated); Status verified 2006-03

CONDITIONS: Kidney Transplant
Keywords: Campath-1H, low-dose immunosuppression, T regulatives cells
MeSH Terms: interventions — Alemtuzumab

INTERVENTIONS:
Drug: Campath-1H

SUMMARY:
During the past 15 years, however, the superior immunosuppressive efficacy of CsA and the well-known toxicity of long-term steroid therapy have prompted trials of steroid withdrawal from renal allograft recipients at various intervals after transplantation. Steroid withdrawal or avoidance must be balanced against the associated risk of precipitating acute allograft rejection. Moreover, with the current immunosuppressive regimens, by 10 years approximately 50% of grafts will have been lost due mainly to chronic rejection or the side-effects of immunosuppressive therapy. Thus, the quest for therapies that might induce specific immune tolerance - ideally via short-term interventions that would target only the pathogenic immune response and leave the protective host immune response unimpaired - has provided a "holy grail" for transplant immunologists.

The humanized IgG monoclonal antibody Campath-1H has been hypothesized to provide enough immunosuppression that would allow maintenance therapy with low-dose CsA, and possibly reprogramming the immune system so to encourage tolerance processes. Despite Campath-1H immunosuppressive regimens have been claimed to induce a condition of "almost tolerance", this has not been proved nor evidence of development of persistent regulatory immune responses long-term post transplant has been provided. Thus, characterizing phenotypically and functionally distinct subsets of T-regulatory cells possibly generated selectively in non-rejecting transplant recipients in Campath-1H-based immunosuppressive regimens may help to find new noninvasive markers of immune system activation to tailor immunosuppressive protocols.

The primary aim of the study is to compare the effect of Campath-1H, low dose sirolimus versus Campath-1H, low dose CsA, both in addition to low dose MMF on phenotypic and functional profiles of peripheral blood mononuclear cells (PBMCs) in kidney transplant recipients in a steroid-free regimen.

DETAILED DESCRIPTION:
The last 40 years have been a period of remarkable evolution of organ transplantation from nothing to a well-established form of treatment with good short-term results. These findings were achieved mainly using the conventional triple-drug regimen with cyclosporine (CsA), azathioprine (or mycophenolate mofetil, MMF), and steroids. During the past 15 years, however, the superior immunosuppressive efficacy of CsA and the well-known toxicity of long-term steroid therapy have prompted trials of steroid withdrawal from renal allograft recipients at various intervals after transplantation, Few transplant centers have also adopted a steroid-free immunosuppressive regimen. Reported benefit of eliminating steroids from immunosuppressive regimens of CsA-treated renal transplant recipients have included improvement of hypertension, hyperlipidemia, glucose intolerance and, in children, acceleration of growth. Avoiding these steroid-related side effects would contribute to improve long-term outcome of the grafts. These and other benefits of steroid withdrawal or avoidance must be balanced against the associated risk of precipitating acute allograft rejection. Moreover, with the current immunosuppressive regimens, by 10 years approximately 50% of grafts will have been lost due mainly to chronic rejection or the side-effects of immunosuppressive therapy. Thus, the quest for therapies that might induce specific immune tolerance - ideally via short-term interventions that would target only the pathogenic immune response and leave the protective host immune response unimpaired - has provided a "holy grail" for transplant immunologists. We now have a number of extremely powerful immunosuppressive drugs and antibodies with different mechanisms of action and the stage is set for a move from current continuous high dose immunosuppressive maintenance therapy to low dose or no maintenance immunosuppression. Indeed, true tolerance can occur in man, examples being successful bone marrow transplantation and patients with liver grafts who have stopped immunosuppression after years of good function.

The humanized IgG monoclonal antibody Campath-1H with a unique target CD52 on T, B lymphocytes and monocytes has been used to eliminate lymphocytes from the blood for more than a month in kidney transplant recipients. Given its potent but safe effect of depleting T and B cells, Campath-1H has been hypothesized to provide enough immunosuppression that would allow maintenance therapy with low-dose CsA, and possibly reprogramming the immune system so to encourage tolerance processes. This has been formally tested in 31 patients undergoing first cadaver renal allograft. The results with a mean two year follow-up have been encouraging, 29 patients having good graft function without receiving maintenance steroids. Similar results have been achieved recently combining Campath-1H and full dose sirolimus in renal transplant recipients. Twenty-three out of 24 patients had good graft function 1 year post transplant. However, most patients were on a lipid-lowering agent to counteract the hyperlipidemic effect of sirolimus. It should be also considered that in both clinical trials acute rejection episodes early post transplant occurred in 20-25% of the patients. Thus, to reduce the risk of hyperlipidemia associated with the current full-dose of sirolimus, while minimizing the risk of rejection, a combination regimen of low dose sirolimus and low dose MMF is worth investigating.

Despite Campath-1H immunosuppressive regimens have been claimed to induce a condition of "almost tolerance", this has not been proved nor evidence of development of persistent regulatory immune responses long-term post transplant has been provided. Thus, characterizing phenotypically and functionally distinct subsets of T-regulatory cells possibly generated selectively in non-rejecting transplant recipients in Campath-1H-based immunosuppressive regimens may help to find new noninvasive markers of immune system activation to tailor immunosuppressive protocols.

Aims of the study

This prospective study in adult kidney transplant recipients is designed with the following aims:

Primary To compare the effect of Campath-1H, low dose sirolimus versus Campath-1H, low dose CsA, both in addition to low dose MMF on phenotypic and functional profiles of peripheral blood mononuclear cells (PBMCs) in kidney transplant recipients in a steroid-free regimen.

Secondary

To compare in the two groups of kidney transplant recipients at 6 and 12 months post-Tx:

* Incidence of acute allograft rejection
* Time course of graft function (as serum creatinine concentration)
* Time course of glomerular filtration rate (GFR)
* Systolic and diastolic blood pressure
* Need for antihypertensive therapy
* Lipid profile (cholesterol, triglycerides, HDL)
* Need for statins
* Fasting blood glucose and need of antidiabetic agents
* 24 h urinary protein excretion rate
* Patient and graft survival
* Incidence of major adverse events (post-transplant anuria, major infections, cancer, abnormal liver function tests, and abnormal hematological blood cell count)

As an extension of the project, patients still on the study at month 12 post-transplant, with no biopsy evidence of acute or chronic rejection, persistent donor specific unresponsiveness and intact 3rd party response in MLR, presence of immune regulatory cells in the peripheral blood will undergo a program of sequential withdrawal of the maintenance low dose immunosuppressive drugs.

Randomization Group 1 (n=11): Campath-1H, low dose sirolimus, low dose MMF These patients will receive Campath-1H at day 0 of transplant. Low dose sirolimus (target to trough concentration of 5-10 ng/ml) and low dose MMF (750 mg twice a day) will be given orally starting on the day of transplant (the first few days through nasogastric tube).

Methylprednisolone (500 mg) will be administered intravenously on day 0, 1, and 2 posttransplant.

The first treatment will be performed 30 min before the dose of Campath-1H, to minimize reactions to cytokine release. Group 2 (n=10): Campath-1H, low dose CsA, low dose MMF The patients will receive Campath-1H at day 0 of transplant. Low dose CsA (target blood C2 level: 450-750 ng/ml) and low dose MMF (750 mg twice a day) will be given orally starting on the day of transplant (the first few days through nasogastric tube). Methylprednisolone will be administered intravenously on day 0 (500 mg), 1 (250 mg), and 2 (125 mg) post-transplant.

The first treatment will be performed 30 min before the dose of Campath-1H, to minimize reactions to cytokine release.

Randomization will be performed at the Clinical Research Center for Rare Disease Aldo eCele Daccò of the Mario Negri Institute for Pharmacological Research.

Study design All patients entering the study will be managed according to standard protocols already in use at the participating Centers.A tissue sample will be taken from the kidney just after harvesting from the donor and, by percutaneous renal biopsy, at the end of the 12 month follow-up for morphological evaluation. Beside conventional histological examination. immunostaining for cytokines, and possible mediators of chronic renal injury (ET-1, TGF-β, RANTES) will be performed. Clinical parameters will be monitored at least every month. Functional parameter will be evaluated at month 6 and 12 post-transplant. Moreover,blood CsA C2, blood sirolimus trough levels, and plasma MMF trough levels will be monitored.

All patients will undergo immunophenotyping of circulating peripheral blood leukocytes at different time points post-transplant. All patients will also undergo lymphocyte function assays at different time points posttransplant.

These assays will be performed pre-transplant, at day 15 and 30 post-transplant (or at the time of acute rejection and after recovery of graft function), at month 6, 12 post-transplant or at the time of any biopsy due to chronic deterioration of graft function and at the time of graft loss.

At the same time points cytokine detection in antigen-activated T cells will be measured by ELISPOT assay.

ELIGIBILITY:
Inclusion Criteria:

* Eligible kidney transplant according to standard criteria
* Recipient of first kidney transplant
* Cadaver or living-related donor
* Written informed consent

Exclusion Criteria:

* Panel reactive antibodies titer >50%
* HLA identical
* High risk of recurrence of renal disease (FSGS, vasculitis, membranous nephropathy)
* Primary and secondary hyperlipidemia
* Platelet count <150000/microliter
* Specific contraindication to the study drug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21
Dates: Start 2003-02; Study Completion 2010-04

PRIMARY OUTCOMES:
Time course of immunophenotyping and lymphocyte function assays in the two groups of kidney transplant recipients randomized to low-dose sirolimus or CsA- based maintenance immunosuppression after Campath-1H induction therapy
Graft function and survival
Safety of induction therapy with Campath-1H and low-dose maintenance immunosuppressive regimen

CONTACTS AND LOCATIONS:
Overall Officials: Norberto Perico, MD, Principal Investigator — Mario Negri Institute for Pharmacological Research
Locations (1):
- Hospital "Ospedali Riuniti" of Bergamo, Bergamo, Italy